CLINICAL TRIAL: NCT02333604
Title: Cancer Experience Registry: An Online Survey Research Study to Understand the Experiences of Cancer Patients and Caregivers
Brief Title: Cancer Experience Registry (CER) for Cancer Patients and Caregivers
Acronym: CER
Status: Recruiting | Type: Observational
Sponsor: Cancer Support Community, Research and Training Institute, Philadelphia (Other)
Responsible Party: Principal Investigator, Erica E. Fortune, Vice President, Research, Cancer Support Community, Cancer Support Community, Research and Training Institute, Philadelphia
Other Study IDs: Salus IRB # 23044
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Neoplasms; Cancer; Caregiver
Keywords: cancer; cancer survivorship; psychosocial needs; cancer experience; acute myelogenous leukemia; breast cancer; breast cancer, metastatic; chronic lymphocytic leukemia; chronic myeloid leukemia; liver cancer; lung cancer; melanoma; multiple myeloma; myelodysplastic syndrome; ovarian cancer; prostate cancer; stomach cancer; bladder cancer; colorectal cancer; patient insights
MeSH Terms: conditions — Neoplasms; Leukemia, Myeloid, Acute; Breast Neoplasms; Neoplasm Metastasis; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Liver Neoplasms; Lung Neoplasms; Melanoma; Multiple Myeloma; Myelodysplastic Syndromes; Ovarian Neoplasms; Prostatic Neoplasms; Stomach Neoplasms; Urinary Bladder Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Cancer Experience Registry®: An Online Survey Research Study to Understand the Experiences of Those Impacted By a Cancer Diagnosis. The Registry is a web-based platform to distribute cross-sectional and longitudinal surveys. Study surveys are designed based on input from advisor experts, including patients and caregivers, and focus on the social, emotional, physical, financial and decision-making experiences of those who have been diagnosed with cancer and their caregivers. Findings contribute toward enhancing care for patients, survivors and caregivers via programming and policy initiatives.

DETAILED DESCRIPTION:
The aims of the Registry are to: 1) better understand the psychosocial experiences and needs of people who have been impacted by cancer, including patients, survivors and caregivers; 2) inform the research community, healthcare providers, patient advocates and policy makers around gaps in care and the psychosocial challenges of people affected by cancer; 3) use the findings to develop and disseminate tailored (data-guided) programs and services that will address the emotional and social needs and ultimately improve the long-term quality of life of people affected by cancer; 4) link registrants to cancer related resources and programs via an online, modifiable platform; and 5) provide collaborating sites (e.g., hospitals/health networks/CSC affiliates) with aggregated reports on quality and needs of members or customers to enhance or improve quality of care.

Findings from the Registry are disseminated online at https://www.cancersupportcommunity.org/sites/default/files/file/2020-07/CSC_Registry_Report_June_2020.pdf

ELIGIBILITY:
Inclusion criteria:

* Have received a cancer diagnosis or have been a family caregiver or informal caregiver (i.e., a relative or friend) for someone diagnosed with cancer
* Live in United States, a US territory, or Canada
* Able to read and understand English

Exclusion criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any individual who has received a cancer diagnosis or has been a family caregiver or informal caregiver for someone diagnosed with cancer
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported quality of life measures | 7 days
  Participant self-reported symptoms and functioning will be measured using the Patient-Reported Outcomes Measurement Information System-Preference Score (PROMIS-Pr). Five domains assess symptoms with higher scores corresponding to worse symptomology (Depression; Anxiety; Pain Interference; Fatigue; Sleep Disturbance) and three assess function with lower scores corresponding to worse functioning (Physical Function; Ability to Participate in Social Roles and Activities; Cognitive Function). Participants rate each item with reference to the past seven days; function scales have no timeframe specified. Scale scores are converted to standardized T scores (mean = 50, SD = 10); normative reference groups are the U.S. general population, except Sleep Disturbance, where comparisons are to a mix of the U.S. population and people with chronic illness.

CONTACTS AND LOCATIONS:
Overall Officials: Erica E. Fortune, PhD, Principal Investigator — Cancer Support Community
Locations (1):
- Cancer Support Community Research & Training Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
IPD is not available at this time. Data in aggregate is shared with recruitment partners.

REFERENCES:
- See also: The 2020 Registry Report highlights findings from the Cancer Experience Registry data — https://www.cancersupportcommunity.org/sites/default/files/file/2020-07/CSC_Registry_Report_June_2020.pdf

DOCUMENTS (1):
  • Informed Consent Form (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT02333604/ICF_004.pdf